CLINICAL TRIAL: NCT04258813
Title: Onco-primary Care Networking to Support TEAM-based Care - the ONE TEAM Study
Brief Title: Onco-primary Care Networking to Support TEAM-based Care
Acronym: ONE TEAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: PRO00104179
Record Dates: First submitted 2020-01-23; First posted 2020-02-06 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Blood Pressure; Hypertension; Cancer; Cancer, Breast; Cancer of Prostate; Cancer Colorectal; Cancer, Endometrial; Cancer of Head and Neck; Non Small Cell Lung Cancer; CVD - Cardiovascular Disease; Diabetes Mellitus; Hypercholesterolemia; Diabetes; Cancer of Esophagus; Cancer of Liver; Cancer, Renal Cell; Cancer of Pancreas; Cancer Ovaries
MeSH Terms: conditions — Hypertension; Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Cardiovascular Diseases; Diabetes Mellitus; Hypercholesterolemia; Esophageal Neoplasms; Liver Neoplasms; Carcinoma, Renal Cell; Pancreatic Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Investigators will use a SMART design with 2 randomizations - at the time of enrollment and after the 12-month measurement. At enrollment, participants will be cluster randomized to the self-guided multi-level iGuide intervention or control arm. An adaptive intervention will be used for the second randomization. PCP clinics in the intervention arm in which 90% or more of their participating patients do not meet the modified HEDIS quality metrics at the 12-month measurement will be considered 'non-responders' and randomized to a tailored/targeted intervention (iGuide2) or a control (iGuide).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): 40 PCP clinics; 400 patients
  Interventions: Behavioral: Control
- iGuide Intervention (Experimental): 40 PCP clinics; 400 patients
  Interventions: Behavioral: iGuide Intervention (Self-guided); Behavioral: iGuide 2 Intervention (Tailored/Targeted)

INTERVENTIONS:
Behavioral: iGuide Intervention (Self-guided) — The iGuide Intervention consists of two patient-level and four PCP-level components. These components include: (1) the patient-level brief video vignettes with a written summary; and (2) patient-facing webinars. The investigators will not use any institutional branding in the videos, printed materials, or recorded webinars so that these deliverables can be used in other settings.
  Arms: iGuide Intervention
Behavioral: iGuide 2 Intervention (Tailored/Targeted) — The iGuide2 patient-level intervention will use a stage-based, tailored approach to four monthly 5-minute video vignettes that incorporates a pre-video worksheet. The investigators will send the worksheets and video vignettes in the method preferred by the patient.
  The targeted iGuide 2 PCP-level intervention will include a cancer specialist-facing dashboard that includes the specialists's patients who are enrolled in the study and are in the intervention arm. The HEDIS quality measures for our three CVD comorbidities will be used. The dashboard will be populated with data available in Epic for the specific patient. If some information is missing (i.e., there is no lipid profile in the laboratory tab), the dashboard will query the PCP via an e-consult, asking to supply the information. Bimonthly, starting with the second randomization, an asynchronous specialist-to-PCP e-consult will be sent to PCPs whose patient(s) do not meet all three of the HEDIS quality metrics.
  Arms: iGuide Intervention
Behavioral: Control — Participants randomized to the control group (n=400) will receive current guideline-concordant cancer care. The investigators will also provide information for healthy living during and after cancer and for preparing for transition from cancer therapy to follow-up care. Monthly, patient education material on healthy living will be sent to the participants via the patient portal or by mail, based on participant preference. At the completion of therapy, they will be provided the NCI Facing Forward:Life After Cancer booklet. Note, this approach is not fully equivalent to an attention control as there will be touch points in the iGuide and iGuide2 interventions that the investigators cannot match for the control group. Also, the research team will not engage the PCPs in clinics randomized to the control group.
  Arms: Control

SUMMARY:
The proposed ONE TEAM Study is an 18-month, cluster randomized controlled trial. This study will use a sequential multiple assignment randomized trial (SMART) design with a second randomization for the intervention group using a dynamic treatment regimen approach. The investigators propose to randomize 800 adults with newly-diagnosed selected cancers treated with curative intent (breast, prostate, colorectal, endometrial, non-small cell lung, and endometrial) and with >1 selected cardiovascular disease (CVD) comorbidity (hypertension, type 2 diabetes mellitus, hypercholesterolemia). Participants will be enrolled through Duke Cancer Institute and two community-based oncology practices, both settings serving socio-demographically diverse populations. The unit of randomization will be the PCP clinic; there will be ~80 PCP clinics across North Carolina involved in the study. The overarching goals of this study are to improve chronic disease management and communication among cancer survivors by engaging PCPs as active members of the cancer care team and reframing the message to cancer survivors and providers.

A diversity supplement with retrospective and qualitative components has been added to abstract older adults with solid tumors who underwent cancer surgery at DUHS. Aims include (1) to estimate the prevalence of cardiovascular complications ≤90 postoperative days among older adults with solid tumors undergoing surgery, and its association with care coordination between surgical providers and PCPs ; (2) to develop a risk index for cardiovascular complications ≤90 days of surgery among older adult patients with a solid tumor; and (3) to Assess experience and perceptions of PCPs on care coordination with surgical providers of older adults with a solid tumor following cancer surgery.

DETAILED DESCRIPTION:
This is an 18-month cluster randomized controlled trial using a SMART design with two randomizations (the second using an embedded dynamic treatment regimen), with a target enrollment of 800 patients with one of six solid tumors (stage I-III breast, prostate, colorectal, endometrial, and head/neck cancer; stage I-II non-small cell lung cancer) who are being treated with curative intent. To engage the PCP early in the process, the investigators will enroll patients at one of their first visits with a cancer specialist (e.g., surgeon, radiation or medical oncologist). The investigators estimate that 80 unique community-based PCP clinics across North Carolina will be involved in the study. The investigators will determine the effectiveness of the multi-level intervention compared with usual care on (1) Healthcare Effectiveness Data and Information Set (HEDIS) quality measures of management of the three CVD comorbidities using laboratory testing (glycated hemoglobin [A1c], lipid profile) and blood pressure measurements; (2) medication adherence assessed pharmacy refill data using Proportion of Days Covered (PDC); and (3) patient-provider communication (Patient-Centered Communication in Cancer Care, PCC-Ca-36).

Key aspects of the intervention are to: reframe the message to patients, PCPs, oncologists, and the respective health care teams in these two settings to emphasize the importance of optimizing the management of comorbidities during and after cancer therapy; promote a change in the workflow in both PCP and oncology practices; enhance PCP-oncologist relationships, and utilize EHR technology. There are two phases of the intervention, both having patient- and PCP-level components. During the first phase of the intervention, occurring with the first randomization, the investigators will test the effectiveness of a self-guided, informational strategy (iGuide). For PCP clinics that do not achieve the HEDIS targets, a booster phase with tailored (patient-level) and targeted (PCP-level) strategies will be tested with a second randomization (iGuide2).

The intervention has been designed to leverage communication tools with in our electronic health record (EHR), Epic . For patients who agree to receive study communications through Epic's patient portal, MyChart, we created an automated messaging system using a dynamic, rules-based protocol which determines the proper language to send each subject based on their study arm and time since enrollment. We developed a similar rules-based automated messaging system for provider communications. This method sends letters to a provider's Epic inbox, called InBasket, for Duke providers and PCPs in the community who have limited access to the Duke EMR through a portal called MedLink. Epic will send letters to PCPs outside of Duke who do not have MedLink access by fax. These outside providers will also be given the opportunity to enroll in MedLink if they are interested.

All participants in the study will be given a survivorship care plan based on the American Society of Clinical Oncology (ASCO) template. Because the investigators will be recruiting participants at our cancer centers and community practices, there will be an inevitable contamination across cancer specialists. Thus, the investigators did not include an oncology-level intervention. However, cancer specialists are integral to the patient- and PCP-level interventions. At the end of the study, patients and PCPs will be mailed a newsletter with a summary of the study findings. Lastly, it is inevitable that some patients will change their PCP during the study. When notified of the change, the research team will send the new PCP the intervention materials.

Supplement:

A retrospective data analysis of Duke cancer registry data integrated with EHR data elements linked by the medical record number will done. The study cohort will consist of older adults ≥65 years who have ≥1 cardiovascular comorbidity (hypertension, type 2 diabetes, dyslipidemia) and underwent cancer surgery for solid tumors at DUHS from January 1st, 2017 to December 31st 2019. Cancers of interest are breast, prostate, colorectal, endometrial, gastric, esophageal, liver, pancreatic, renal cell, bladder, ovarian, head/neck, and non-small cell lung cancer. Cancer diagnoses will be grouped according to the International Classification of Diseases for Oncology, 3rd revision (ICD-O-3). Key variables to be abstracted include demographic, clinical (comorbidities & pertinent history, medications, cancer treatment, labs), geriatric-specific (frailty, function, cognition, operative, post-operative, and PCP follow-up data.

The qualitative component will involve semi-structured interviews with PCPs of older adults with solid tumors who underwent cancer surgery within a 12-month period in the DUHS. Participating PCPs will complete an audio-recorded semi-structured interview that will last approximately 30 minutes. Qualitative interview: We will design a semi-structured interview guide assessing perspectives on (1) frequency, modes, and perceived quality of communication with surgical providers during transitions in care from surgery (2) perceived barriers to effective care coordination with surgical providers (3) how communication and care coordination can be improved. Open-ended prompts may include "Please describe your experience with care coordination with surgical providers of older adults undergoing cancer surgery?" "What challenges have you faced when communicating with surgical providers of your older adult patients?"; "What are your thoughts on ways to improve communication and care coordination after an older adult with solid tumor undergoes surgery?", "Please give examples of particularly good or poor care coordination with surgical providers?" The interview guide will be designed with assistance from the experienced research staff in the Duke Behavioral Health and Survey Research Core.

Power re-estimation:

Our original power calculations were completed using methods described in Eldridge et al (ref). At the time of project development, the number of practices (40 per arm) and number of patients per practice (10) were unknown, but we estimated the 10 when computing planned sample size for the study. Following enrollment patterns over time, it has been determined that the average number of patients per practice is much smaller, 1.81, presently. If we had this information at time of study planning, based on the design effect and our original effect size, we see that with smaller sample size than originally planned/proposed, we still retain high power, primarily due to the reduction in the design effect (DE). Using the revised calculations, we estimate a power of 0.85-0.9 for 250 projected randomized participants and a power of 0.9 for 275 projected randomized participants.

ELIGIBILITY:
Inclusion Criteria:

A total of 800 individuals who fall under the following criteria will be enrolled:

* Diagnosed with -

  * Stage I-III breast [female], colorectal, endometrial (carcinomas), head/neck [H/N] and non-small cell lung cancer [NSCLC]
  * Stage I-IV prostate cancer
  * Organ transplant recipients are not excluded as long as kidney function is within eligible range
  * Chronic Lymphocytic Leukemia or small lymphocytic lymphoma on first or second line treatment
* Treated with curative intent (not applicable for patients diagnosed with CLL/SLL)
* 18-79 years old
* Has at least one of three CVD comorbidities (hypertension, diabetes, or hypercholesterolemia) - based upon whether the patient is currently on a medication for the comorbidity at time of recruitment
* Had a visit with their PCP in the previous 12 months

Patients will be approached for study participation within 120 days of starting their cancer treatment at Duke (except for men with prostate cancer on androgen deprivation therapy [ADT] and those previously on active surveillance). Those coming off active surveillance to receive treatment will be approached within the next 120 days. Men with prostate cancer that are on ADT can be approached for consent at any time while on treatment.

Supplement:

A sample size of 2800-3000 patients will be pulled from the Duke Cancer Registry. The retrospective cohort will consist of older adults ≥65 years who have ≥1 CVD comorbidity (hypertension, type 2 diabetes, dyslipidemia) and underwent cancer surgery for solid tumors (breast, prostate, colorectal, endometrial, gastric, esophageal, liver, pancreatic, renal cell, bladder, ovarian, head/neck, and non-small cell lung cancer) at DUHS from January 1st, 2017 to December 31st 2019.

The qualitative component of the supplement (Appendix IV: Aim 3) will involve 12-20 PCPs who arepart of the Duke Primary Care Research Consortium. Eligible PCP participants will be English-speaking providers who have provided care to ≥1 older adult patient who has undergone cancer surgery within a 12-month period at DUHS.

Exclusion Criteria:

Individuals with a history of the following conditions will be ineligible:

* Myocardial infarction in the previous 24 months
* Stage III-IV heart failure (EF <30%)
* Stage IV-V chronic kidney disease (eGFR <30)
* Neuroendocrine tumors
* Uterine sarcomas
* Bilateral axillary dissections - due to the inability to collect an upper extremity BP

Patients who are coming to Duke for surgery only and not planning to return are ineligible. Patients who cannot read, are blind or do not understand/speak English will not be enrolled.

Participants who progress to metastatic disease during the course of the 18-month study period will be allowed to continue to participate unless they voluntarily withdraw from the study.

Additional health information may be assessed on a case by case basis by the PI to determine if the individual is an appropriate candidate for the intervention.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
HEDIS quality measure of management hypertension | 18 months
  BP<140/90 mmHg. Rather than use vital sign BP readings, which tend to have much variation, the research staff will measure the BP at the above time periods. The investigators will assess BP consistent with the TRUE Consortium standards.
HEDIS quality measure of management of diabetes | 18 months
  A1c<8.0%. To evaluate diabetes management, the research team will measure fasting laboratory A1c at the time of each study assessment.
HEDIS quality measure of management of statin use | 18 months
  Statin use if patient is diabetic or has a 10-year ASCVD risk >10%. To evaluate statin use, the research team will measure fasting laboratory lipid profile at the time of each study assessment.
Patient-Centered Communication in Cancer Care | 18 months
  Patient-reported Patient-Centered Communication in Cancer Care (PCC-Ca-36). The PCC-Ca-36 is a 36-item survey that measures one overall communication score, and six sub-domains that are consistent with our conceptual models:exchanging information, making decisions,fostering healing relationships, enabling patient self-management, managing uncertainty, and responding to emotions.
Medication adherence | 18 months
  Medication adherence will be measured as proportion of days covered, and the research team will obtain pharmacy refill data from the EHR. For participants followed by a Duke PCP, all refills (including refill date, amount, number of refills) are captured in Epic. For PCPs outside of Duke, the research team will use the Epic link with Surescripts which captures e-prescribed medications. Using this data, the investigators will calculate the PDC for an index medication from each medication class for the three CVD comorbidities, depending upon the number of CVD comorbidities a participant has. PDC is a measure of how many days a patient is in possession of their medication, calculated as the total number of days in a followup period divided by the total number of days that a medication was available (ratio of the number of days the patient is covered by a medication during a refill period).
Diversity supplement primary outcome: 90-day postoperative cardiovascular complications | 90 days
  any occurrence of myocardial infarction, stroke, venous thromboembolism (deep venous thrombosis, pulmonary embolism), new-onset atrial fibrillation, heart failure or cardiopulmonary arrest within 90 days of surgery tracked with ICD codes.

SECONDARY OUTCOMES:
Medication adherence defined through patient self-report | 18 months
  The investigators will use a self-report adherence measure created and validated by Voils et al which assesses extent of non-adherence as well as reasons for non-adherence. Participants will first respond to adherence items for each CVD comorbidity (n = 3 items each). Participants who are identified as non-adherent will be asked a series of medication-specific reasons for nonadherence (up to 18 items).
Clinical laboratory values | 18 months
  Comparison of A1c levels
Clinical laboratory values | 18 months
  Comparison of LDL-cholesterol levels
Patient activation | 18 months
  Patient activation will be assessed using the Patient Activation Measure (PAM), which is a 13-item measure that assesses a patient's knowledge, skills, and confidence that are central to managing health and health care. The PAM categorizes patients into four levels of activation: disengaged and overwhelmed (level 1), becoming aware but still struggling level 2), taking action (level 3), and maintaining behaviors and pushing further (level 4).
Financial burden | 18 months
  Patients' experience with cost of care (financial burden and objective cost) will be assessed through two self-reported measures of financial burden and actual expenditures. To assess financial burden, or financial toxicity, the research team will collect the Functional Assessment of Chronic Illness Therapy COmprehensive Score for financial Toxicity (COST). The FACIT-COST is an 11-item measure. The research team will also objectively ask patients about the amount of out-of-pocket expenditures for care over the last month via survey questions (e.g., insurance premiums, copayments, prescription medications, etc).
Patient-reported care coordination | 18 months
  Patient-reported care coordination will be collected using a 36-item measure developed by Haggerty et al. The measure contains 9 subscales that address team relational continuity, problems with coordination, gaps in information transfer, and patient's partnership in care.
Provider-reported care coordination | 18 months
  Provider-reported care coordination will be measured using companion clinician-reported measures, the Coordination of Specialty Care - Specialist Survey (n=13 items) and the Coordination of Specialty Care - Primary Care Survey (n=24 items). Both measures were developed by Vimalananda and colleagues, and include companion domains that facilitate descriptive comparisons across measures.The specialist version includes four domains (i.e., Relationships, Roles and Responsibilities,Communication, Data Transfer). The Roles and Responsibilities domain is broken into three domains in the primary care version (i.e., Role Clarity, Communication, Role Agreement, Making Referrals), resulting in a total of 6 factors.

OTHER OUTCOMES:
Risk index for cardiovascular complications | 90 days
  Risk index for cardiovascular complications ≤90 days of surgery among older adult patients with a solid tumor
PCP-reported care coordination | 12 months
  PCPs who are participating in either the intervention or control arms of the ONE TEAM study will be invited to participate in a qualitative semi-structured interview guide assessing perspectives on (1) frequency, modes, and perceived quality of communication with surgical providers during transitions in care from surgery (2) perceived barriers to effective care coordination with surgical providers (3) how communication and care coordination can be improved.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zullig LL, Shahsahebi M, Neely B, Hyslop T, Avecilla RAV, Griffin BM, Clayton-Stiglbauer K, Coles T, Owen L, Reeve BB, Shah K, Shelby RA, Sutton L, Dinan MA, Zafar SY, Shah NP, Dent S, Oeffinger KC. Low-touch, team-based care for co-morbidity management in cancer patients: the ONE TEAM randomized controlled trial. BMC Fam Pract. 2021 Nov 18;22(1):234. doi: 10.1186/s12875-021-01569-8. PMID 34794388

DOCUMENTS (1):
  • Informed Consent Form (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT04258813/ICF_000.pdf